CLINICAL TRIAL: NCT01039909
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Clinical Study to Assess the Effects of SRT2104 Upon Immobilization-Induced Skeletal Muscle Atrophy in Healthy Human Volunteers
Brief Title: A Clinical Study to Assess the Effects of SRT2104 Upon Immobilization-Induced Skeletal Muscle Atrophy in Healthy Human Volunteers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Subjects were never screened/enrolled
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: E.D. Derilus; Clinical Disclosure Advisor, GSK Clinical Disclosure
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 113682; SRT-2104-003; SIR113682
Record Dates: First submitted 2009-12-23; First posted 2009-12-25 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Healthy Volunteer; Atrophy, Muscular
MeSH Terms: conditions — Muscular Atrophy | interventions — SRT2104

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): The Placebo treatment group will be administered 8 placebo capsules per day. Placebo will be administered orally once daily for twenty-eight consecutive days.
  During the clinic visits, the subjects will receive placebo approximately 15 minutes following the start of consumption of a standardized meal. During non-clinic days, the subject will self-administer the test material approximately 15 minutes following the start of consumption of a standardized meal. Test material should be administered with approximately 400 mL of water at approximately the same time every dosing day. Subjects must wait at least 2 hours before consuming additional calories.
  Interventions: Drug: Placebo
- 2.0g SRT2104 (Active Comparator): The 2.0g SRT2104 treatment group will be administered 8 SRT2104 0.25g capsules per day. 2.0g SRT2104 will be administered orally once daily for twenty-eight consecutive days.
  During the clinic visits, the subjects will receive SRT2104 approximately 15 minutes following the start of consumption of a standardized meal. During non-clinic days, the subject will self-administer the test material approximately 15 minutes following the start of consumption of a standardized meal. Test material should be administered with approximately 400 mL of water at approximately the same time every dosing day. Subjects must wait at least 2 hours before consuming additional calories.
  Interventions: Drug: SRT2104

INTERVENTIONS:
Drug: Placebo — For the placebo product, SRT2104 drug substance will be replaced by microcrystalline cellulose (Avicel® PH 105) to match the SRT2104 investigational product.
  Eight size 00 Swedish orange opaque hard gelatin capsules containing placebo are stored in a dosing bottle and provided to all participating subjects for oral ingestion.
  Arms: Placebo
Drug: SRT2104 — SRT2104 investigational product is a size 00 Swedish Orange opaque hard gelatin capsule containing 0.25 g of SRT2104, a new chemical entity which is supplied as a micronized, yellowish/amber powder. Eight SRT2104 capsules are stored in a dosing bottle and provided to all participating subjects for oral ingestion.
  Arms: 2.0g SRT2104

SUMMARY:
The main purpose of this study is to investigate the effect of SRT2104 upon energy production in muscle (specifically the maximum amount of energy produced with muscle contraction), how much sugar and fat are stored in the muscle, and the size of the muscle after receiving 2.0 g of SRT2104 or placebo given in capsule form once a day for 28 days including a 14 day knee and lower leg immobilisation period during the final 14 days of dosing.

Imaging methods, muscle biopsies and exercise tests will be used in the study to see whether the following measurements change after taking SRT2104 for 28 days, including an immobilised knee and lower leg for the final 14 days of dosing.

i) energy reaching the muscles ii) muscle strength iii) changes in the structure of the muscle

This study will also investigate the pharmacokinetics, safety and tolerability of 2.0 g of SRT2104 administered orally once daily for 28 consecutive days. The investigation of pharmacokinetics of SRT2104 allows us to gather information regarding:

i) how long it takes for the drug to be absorbed and detected in the blood ii) how much we can detect iii) how long we can detect it for iv) how often we need to give the drug to maintain a steady amount in the blood.

SRT2104 will be given to healthy subjects aged between 18 and 40 years old. Subjects will participate in this single centre study for approximately 79 days. The study consists of 11 outpatient clinic visits and 4 telephone calls (including a prescreen call to determine whether subjects are interested in participating).

DETAILED DESCRIPTION:
Participants will take part in a prospective, single center, randomized, double-blind, clinical study of 2.0 g/day of SRT2104 or placebo (test material) administered orally as 0.25 g capsules. The study will evaluate the effect of 28 days of consecutive SRT2104 dosing upon muscle strength, metabolism and structure of the ankle muscle group following a 14 day leg immobilization period. The study will also evaluate pharmacokinetic parameters as well as the safety and tolerability of 2.0 g/day of SRT2104. Thirty-four (34) healthy male and female subjects aged 18-40, who fulfill the inclusion/exclusion criteria, will be enrolled in this study. Subjects will be randomized 1:1 to receive either 2.0 g/day of SRT2104 or placebo in a fed state for 28 consecutive days. Subjects will remain on a fixed dose of test material for all dosing days in the study.

Subjects will provide written informed consent and undergo screening assessments. If eligible and willing to participate, subjects will undergo baseline strength testing, muscle biopsy, MRI, and MRS evaluations on Day -1 to assess muscle strength, and metabolism. Participants will then commence a 28 day dosing period with test material. On the first day of dosing (Day 1), pharmacokinetic and safety assessments will be performed. On Day 15, after subjects have completed 14 days of dosing with test material, participants will repeat the muscle biopsy, strength testing, MRI evaluations, pharmacokinetic and safety assessments. Following the study assessments on Day 15, subjects will commence a 14 day immobilization period. The leg of the dominant leg will be immobilized with a temporary removable brace, and subjects will be instructed to ambulate using crutches for the duration of the immobilization period. Designated site staff will contact subjects via telephone on Day 18 and Day 24 to check on the subjects' wellbeing and ability to function while immobilized. Subjects will report to the study site on Day 21 during the 14 day immobilization period for assessment of the immobilized leg, including safety evaluations. On Day 28, following completion of the 14 day immobilization period, a muscle biopsy, skeletal muscle evaluations, pharmacokinetic and safety assessments will be performed. Subjects will return to the clinic for an End of Study visit 7 days (+/- 2 days) after the last dose of test material for follow up safety assessments. A follow-up safety call will be made to each subject approximately 30 days following their final dose of SRT2104 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subjects may be of any race and gender within the age range of 18 to 40 years inclusive
* All female subjects must be of non-childbearing potential. For the purposes of this study, this is defined as the subject being amenorrheic for at least 12 consecutive months, or at least 6 weeks post-surgical bilateral oophorectomy with or without hysterectomy, or women who underwent tubal ligation. For women in menopause, menopausal status will be confirmed by demonstrating levels of follicle stimulating hormone (FSH) 40 - 138 mIU/ml and oestradiol < 20 pg/ml at entry, unless this information is available in the subject's medical record. In the event a subject's menopause status has been clearly established (for example, the subject indicates she has been amenorrheic for 10 years), but FSH and/or oestradiol levels are not consistent with a post-menopausal condition, determination of subject eligibility will be at the discretion of the principal investigator following consultation with the sponsor and Medical Monitor
* All male subjects and their partners must agree to use double-barrier birth control or abstinence while participating in the study and for 12 weeks following the last dose of study drug
* Comprehension of the nature and purpose of the study and compliance with the requirement of the entire protocol
* Willingness and ability to provide written informed consent to participate in the study
* Subject is not taking any concomitant medications which may be associated with thrombosis (e.g., estrogens)
* Have a normal 12-lead ECG or one with changes considered to be clinically insignificant on medical review. QTc must be ≤430msec for males and ≤450msec for females
* No prior history of disease markers for hepatitis B and C virus
* Body Mass Index (BMI) 18-32 kg/m^2 (inclusive)
* Non-smoking status as verified by urinary cotinine levels below 500ng/mL at the screening visit. This can include ex-smokers who have given up smoking for >5 years.
* Absence of significant disease or clinically significant abnormal laboratory values on the laboratory evaluations, medical history or physical examination during screening; normal end organ function, as determined by the Principal Investigator
* Ability to communicate in person and by telephone in a manner that allows all protocol procedures to be carried out safely and reliably in the opinion of the investigative site staff
* Ability to swallow 8 capsules of study medication with 400 mL of water

Exclusion Criteria:

* Any major illness in the past three months or any ongoing chronic medical illness which in the opinion of the PI or Medical Monitor could risk subject safety or interpretation of the results
* History of congenital or acquired coagulopathy, including a history of prior venous thrombophlebitis/thromboembolism
* Family history of hypercoagulable state
* History of bleeding diathesis
* Use of anti-platelet agents other than low dose aspirin, (81 mg per day or equivalent) and/or anti-coagulant medications
* Any condition leading to venous stasis, such as varicose veins or congestive heart failure
* Any surgery of the lower extremity during the last 6 months, except for simple excisions of skin lesions
* Air or other confined travel in excess of two hours within the week prior to enrolment or anticipated at anytime during the study
* History of cancer except non-metastatic, non-melanoma skin cancer or carcinoma-in-situ
* History of renal or liver impairment, including nephrotic syndrome
* Presence of pedal edema
* History of gastro-intestinal surgery or has a current gastrointestinal disease which may influence drug absorption
* History, within 3 years, of drug abuse (including benzodiazepines, opioids, amphetamine, cocaine, and THC) or a positive drug result at the screening visit
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of Screening
* A positive test for HIV antibody
* History of alcoholism, and/or is currently drinking more than two drinks per day on a regular basis (one glass of wine, half a pint of beer, one measure of a spirit)
* Participation in a clinical trial within the past three months (defined as three months from the date of last dose of an investigational medicinal product)
* History of difficulty in donating blood or accessibility of veins in left or right arm
* Blood donation (one unit or 350 mL) within one month prior to receiving test material
* Use of herbal products, over-the-counter medication or prescription drug therapy for which 5 times the half-life is longer than 21 days (i.e., the screening Period) prior to enrolment into the study. Subjects must also refrain from taking herbal products for the duration of the study
* History of a significant physical injury in the past 6 months that resulted in immobilization, impaired ambulation or abnormal range of motion
* History of neuromuscular disease
* A positive pre-study drug/alcohol screen
* A documented history of claustrophobia and/or in vivo ferrous material which will interfere with magnetic resonance examinations
* Subject is exercising more than 30 minutes per session twice weekly

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2011-02 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
To investigate the effect of SRT2104 upon muscle metabolism, specifically mitochondrial function using P31 Magnetic Resonance Spectroscopy following a 14 day leg immobilization within a 28 day SRT2104 dosing period. | Muscle metabolism, specifically mitochondrial function using P31 Magnetic Resonance, will be assessed on Day -1, Day 15 and Day 28.

SECONDARY OUTCOMES:
To investigate muscle metabolism, intra-muscular lipid and glycogen following a 14 day leg immobilization within a 28 day SRT2104 dosing period. | Muscle metabolism, intra-muscular lipid and glycogen will be assessed on Day -1, Day 15, and Day 28.
To investigate the effect of SRT2104 upon muscle strength following a 14 day leg immobilization within a 28 day SRT2104 dosing period. | Muscle Strength is assessed on Day -1, Day 15, and Day 28.
To investigate the effect of SRT2104 upon muscle structure (total muscle volume and muscle structure) following a 14 day leg immobilization within a 28 day SRT2104 dosing period. | Muscle Structure will be assessed on Day -1, Day 15, and Day 28.
To characterize the pharmacokinetic profile of SRT2104 after a single dose and after multiple administrations of SRT2104. | PK samples will be collected on Day1 at pre-dose, 1, 3, 4, 8, and 24hrs post-dose (Day 2). On Day 15 and Day 28, PK samples will be collected at pre-dose, 1, 3, 4, and 24hrs post-dose (Day 16 and Day 29).
To assess the safety and tolerability of 2.0 g/day SRT2104 administered orally for a 28 day dosing period. | For the duration of the study AEs and clinically significant abnormal laboratory values will be recorded based upon investigator observation and subject reporting through a subject diary. Safety will be monitored by AEs, VS, physical exam, labs and ECGs.
To investigate the effect of 14 day administration of SRT2104, using the above mentioned primary and secondary analyses, on normal/mobile muscle function. | Normal/mobile muscle function will be assessed on Day -1, Day 15, and Day 28.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline